CLINICAL TRIAL: NCT05629598
Title: A Phase Ⅱ Clinical Study on the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Polyethylene Glycol Recombinant Human Erythropoietin Injection (CHO Cell) in Optimal Dose and Administration Regimen for Maintenance Therapy in Patients With Regular Dialysis Renal Anemia.
Brief Title: A Study of PEG-EPO Injection (CHO Cells) for Maintenance Therapy of Patients With Renal Anemia .
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Angde Biotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD-006-02
Record Dates: First submitted 2022-06-27; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Renal Anemia
Keywords: PEG-EPO

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A1 (Experimental): Recombinant human erythropoietin injection; Weekly dose of short-acting EPO (IU/kg)* 0.004 (conversion coefficient), Q2W for administration.
  Interventions: Biological: Recombinant human erythropoietin injection
- B1 (Experimental): Recombinant human erythropoietin injection; Weekly dose of short-acting EPO (IU/kg)* 0.008 (conversion coefficient), Q2W for administration.
  Interventions: Biological: Recombinant human erythropoietin injection
- A2 (Experimental): Recombinant human erythropoietin injection; Weekly dose of short-acting EPO (IU/kg)* 0.004 (conversion coefficient), Q4W for administration.
  Interventions: Biological: Recombinant human erythropoietin injection
- B2 (Experimental): Recombinant human erythropoietin injection; Weekly dose of short-acting EPO (IU/kg)* 0.008 (conversion coefficient), Q4W for administration.
  Interventions: Biological: Recombinant human erythropoietin injection
- C (Active Comparator): Human erythropoietin injection；Refer to the product instructions.
  Interventions: Biological: Human erythropoietin injection

INTERVENTIONS:
Biological: Recombinant human erythropoietin injection — The dose of PEG-EPO (CHO cells) is converted according to the average weekly dose of short-acting EPO before randomization (4 weeks before randomization) multiplied by the corresponding conversion coefficient (low conversion coefficient is 0.004, High conversion coefficient is 0.008).
  Arms: A1; A2; B1; B2
Biological: Human erythropoietin injection — Refer to the product instructions
  Arms: C

SUMMARY:
The purpose of the study is to explore the optimal dose and administration of the experimental drug, and to evaluate the safety and efficacy of the drug in patients with renal anemia. Patients with renal anemia on regular dialysis treatment are expected to be enrolled in this study.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open-label, positive controlled phase II clinical study. A total of 125 to 150 patients with renal anemia receiving regular dialysis were enrolled in this study. Those patients were randomly allocated to 5 treatment groups in a ratio of 1:1:1:1:1, with 25 to 30 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients at the age of 18~75 (including critical value).
2. Patients clinically diagnosed with renal anemia who have received dialysis for at least 12 weeks (hemodialysis≥3 times/week, total urea clearance index (Kt/V) ≥1.2 or urea reduction rate (URR) ≥65%; peritoneal dialysis≥4 times/day, weekly Kt/V≥1.7);
3. Hb in screening period should be within the range of 100~130g/L (including both ends), and the deviation should not exceed 10g/L;
4. Iron status (TSAT ≥20% or SF ferritin ≥100μg/L) during screening.
5. Have been stably treated with short-acting EPO 1-3 times per week for at least 12 weeks before baseline;
6. Consent to use reliable contraceptive methods and no family planning from the screening period to 3 months after the last administration；
7. Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Patients with a history of severe allergies (including drug allergies), especially allergic to erythropoietin, or to any component of the test drug (e.g. polyethylene glycol);
2. Have a history of kidney transplantation or plan to undergo kidney transplantation during the trial；
3. Have any other disease that causes chronic anemia (e.g., sickle cell anemia, myelodysplastic syndrome, hematologic malignancy, myeloma, hemolytic anemia, pure red cell aplastic anemia) or PRCA following therapy of erythropoietin protein;
4. Suffered from acute or chronic blood loss (such as gastrointestinal bleeding) or undergwent surgical procedures due to massive bleeding within 3 months before screening, or plan to have a surgery during the clinical trial (except for arteriovenous fistula or peritoneal dialysis tube adjustment);
5. Have a history of malignant tumors within the past 5 years (excluding non-melanoma skin cancer or excised carcinoma in situ);
6. Suffer from autoimmune diseases (such as rheumatoid arthritis or systemic lupus erythematosus) or diseases of endocrine system (such as poorly controlled diabetes mellitus complicated with peripheral vascular diseases, severe secondary hyperparathyroidism [parathyroid hormone > 800ng/L]);
7. Received systemic antibiotic treatment or C-reactive protein ≥30mg/L within 4 weeks due to severe infection before screening;
8. The following conditions occur during screening period:

   Hepatic dysfunction (AST or ALT>3 times ULN); Coagulation dysfunction (activated partial thrombin time > 1.5 times ULN); Folic acid or vitamin B12 deficiency (serum folic acid level <LLN, vitamin B12 <LLN); Positive for HBsAg, HBcAb, HIV-ABb, HCV-AbB or TP-Ab;
9. Suffer from severe thromboembolic disease, poorly controlled severe hypertension (SBP before dialysis > 170mmHg or DBP ≥100mmHg) or hypotension (SBP before dialysis <90mmHg);
10. Suffer from severe cardiovascular and cerebrovascular disease, severe or unstable coronary artery disease, heart failure (NYHA CLASS III or IV), or those who received coronary artery bypass grafting or percutaneous coronary intervention within 6 months, or those who had a history of myocardial infarction or stroke within 3 months;
11. Received androgen therapy or blood transfusion within 8 weeks before screening period;
12. Received long-acting ESAs within 3 months or HIF-PHI (e.g., rosalat) within 2 weeks before initial administration;
13. Participated in other clinical trials as a subject within 4 weeks before screening period or the duration from the last administration to enrollment was shorter than the 5 half-lives of the drug;
14. Have a history of epileptic seizures or mental illness;
15. Alcoholism, drug abuse or drug addiction
16. Pregnant or breastfeeding;
17. Investigator considers not suitable to enter this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-03-17 (Estimated); Study Completion 2023-08-16 (Estimated)

PRIMARY OUTCOMES:
Change of mean hemoglobin compared to baseline during fixed treatment | Day1-Day42
  Change of mean hemoglobin (Hb) content from baseline during fixed treatment (fixed treatment：week 1 to week 6)
Change of mean hemoglobin during dose adjustment period | Day85-Day126
  Change of mean hemoglobin compared to baseline from week 13 to 18 during dose adjustment period (dose adjustment period: week 7 to week 18/week 20).

SECONDARY OUTCOMES:
Proportion of patients with hemoglobin keeping within the target range | Day1-Day42、Day85-Day126
  Proportion of patients with hemoglobin keeping within the target range (target range: the variation from baseline Hb is within ±10g/L, and HB is in the range of 100-130g/L) during treatment period (fixed treatment, week 13 to 18 during dose adjustment period).
Reticulocyte count, Hematocrit, Erythrocyte count | Day1-Day42、Day85-Day126
  Changes of mean values of other evaluation indexes (including HCT, RET, RBC) between baseline and different stages of treatment (fixed treatment period, week 13 to 18 of dose adjustment period).
Proportion of patients receiving red blood cell transfusion and number of transfusions during the trial. | Day1-Day126/140
Number of iron deficiency, number of patients and proportion of patients with iron deficiency during the trial | Day1-Day126/140
  Iron deficiency was defined as SF≤100μg/L and TSAT≤20% in peritoneal dialysis subjects; SF≤200μg/L and TSAT≤20% in hemodialysis subjects.
The number and proportion of patients with dose adjustments during the trial | Day1-Day126/140
Anti-drug antibody | 1,5, 9, 13, 17 weeks (before administration) and 28±2 days after the last administration (A2/B2group ,A1/B1 patients with intensive blood collection) or 14±2 days after the last administration (A1/B1 patients with sparse blood collection)
  The incidence of ADA and Nab
Adverse events | Day1-Day126/140
  Any adverse event that occurred during the clinical trials of all patients.
Cmax | Day1-Day126/140
  Maximum observed plasma concentration of EPO.
Tmax | Day1-Day126/140
  Time to maximum observed plasma concentration of EPO.
AUC 0-t | Day1-Day126/140
  Area under the plasma concentration-time curve from time 0 to the time of the last measurable concentration of EPO.
AUC 0-∞ | Day1-Day126/140
  Area under the plasma concentration-time curve from time 0 to infinity.
Emax | Day1-Day126/140
  Maximal effect concentriation
Tmax of Emax | Day1-Day126/140
  Time to maximal effect concentriation
AUE0-t | Day1-Day126/140
  Area under the plasma effect-concentriation curve from time 0 to the time of the last measurable concentration of EPO.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospitial,College of Medicine,Zhejiang University, Hanzhou, Zhejiang, China